CLINICAL TRIAL: NCT01158417
Title: Effect of Resveratrol on Insulin Resistance and Inflammatory Mediators in Obese and Type 2 Diabetic Subjects
Brief Title: Resveratrol in Type2 Diabetes and Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA clinical hold requiring IND submission, product not available in the market anymore
Sponsor: University at Buffalo (Other)
Collaborators: Kaleida Health (Other)
Responsible Party: Principal Investigator, Paresh Dandona, MD, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1935
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Type 2 Diabetes; Obesity; Insulin Resistance
Keywords: Type 2 Diabetes; Obesity; Insulin Resistance; Resveratrol; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Insulin Resistance; Inflammation | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo
- Resveratrol 40 mg oral three times a day (Experimental): Resveratrol
  Interventions: Drug: Resveratrol 40 mg oral three times a day
- resveratrol 500 mg oral once daily. (Experimental): Resveratrol
  Interventions: Drug: Resveratrol 500 mg oral once daily.

INTERVENTIONS:
Drug: Placebo — oral
  Arms: Placebo
Drug: Resveratrol 40 mg oral three times a day — Drug
  Other Names: Resveratrol 40mg
  Arms: Resveratrol 40 mg oral three times a day
Drug: Resveratrol 500 mg oral once daily. — Resveratrol 500 mg oral once daily.
  Other Names: Resveratrol 500 mg
  Arms: resveratrol 500 mg oral once daily.

SUMMARY:
The main objective of this study is to investigate the effect of resveratrol (plant derived food supplement) on inflammatory mediators and insulin resistance at the cellular and molecular level in obese non diabetic and type 2 diabetic subjects in vivo.

DETAILED DESCRIPTION:
The main objective of this study is to investigate the effect of resveratrol on inflammatory mediators and insulin resistance at the cellular and molecular level in obese non diabetic and type 2 diabetic subjects in vivo. This research will investigate the hypothesis that resveratrol, when given orally to obese and type 2 diabetic subjects induces a decrease in reactive oxygen species (ROS) generation and the pro-inflammatory transcription factor nuclear factor-kB (NF-kB) and the inflammatory mediators regulated by it. The hypothesis that resveratrol suppresses the high fat, high carbohydrate (HFHC) meal induced inflammatory and oxidative response, will also be investigated. This research will also investigate the hypothesis that resveratrol intake for 12 weeks improves insulin sensitivity by lowering the Homeostasis model assessment of insulin resistance (HOMA-IR), an index of insulin resistance and, that resveratrol intake will cause an increase in incretins.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years of age and older
2. Healthy Obese subjects with BMI > 30
3. Type 2 Diabetics with BMI > 30
4. Subjects with good peripheral vein.
5. Subjects on statins, ACE inhibitors and thiazolidenediones will be allowed as long as they are on stable doses of these compounds and the dosage is not changed during the course of study.

Exclusion Criteria:

1. Subjects on any antioxidant medication
2. Patient on non-steroidal anti-inflammatory drug
3. On any agent with significant antioxidant properties.
4. History of drug or alcohol abuse
5. Any life threatening disease
6. Allergy to peanuts, grapes, wine, mulberries.
7. Pregnant women.
8. Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass surgery or coronary angioplasty) in the previous four weeks.
9. Subjects on anticoagulants.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2012-07-08 (Actual); Study Completion 2012-07-08 (Actual)

PRIMARY OUTCOMES:
NF-Kb | 12 weeks
  To investigate the effect of resveratrol on ROS generation and the pro-inflammatory transcription factor NF-kB

SECONDARY OUTCOMES:
GLP-1 | 12 weeks
  To see whether Resveratrol leads to a greater stimulation of the incretin system and secretion/release of GIP and GLP-1 when compared to that following placebo

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, Principal Investigator — Kaleida Health
Locations (1):
- Jeanne Hejna, Williamsville, New York, United States